CLINICAL TRIAL: NCT06866210
Title: Analyse Du Risque De Rupture Des AnévrysMes Intracrâniens Au Travers Des Déterminants Sociaux De Santé
Brief Title: Risk Analysis of Intracranial Aneurysm Rupture Through Social Determinants of Health
Acronym: ARAMISS
Status: Active, not recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0009; DAtAE-2023-5 (Other Grant/Funding Number: DGOS)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Social Determinant of Health; Intracranial Aneurysms; Subarachnoid Hemorrhage; Treatment Outcomes; Natural Languages Processing; Observational Study; Aneurysm, Ruptured
Keywords: Social Determinant of health; Intracranial aneurysm; Subarachnoid hemorrhage; Treatment Outcomes; Natural languages processing; Observational study; Epidemiology; Data warehouse
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage; Aneurysm, Ruptured

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ruptured IA or unruptured IA: ruptured IA or unruptured IA

SUMMARY:
Intracranial aneurysms (IA) are arterial malformations affecting about 3% of the overall population. Rupture is the most severe complication, as it is associated with nearly 30% of death or severe disability. The available scores to assess rupture risk are mainly based on usual modifiable and non-modifiable risk factors from the literature, but they appear insufficient to predict rupture. Emerging factors, such as sleep apnea syndrome and the use of certain medications, seem to influence the risk of rupture. The study of social determinants of health (SDOH) is highly relevant, given numerous reports showing the impact of SDOH, in addition to vascular risk factors, on vascular diseases like ischemic stroke or myocardial infarction.

It is therefore reasonable to study the interaction between rupture risk factors and SDOH on the rupture risk of IA. Several initiatives have been undertaken to assess rupture risk, but few have included SDH. Limitations were often raised, especially regarding data accessibility. However, it is now possible, thanks to artificial intelligence (AI) algorithms, particularly natural language processing (NLP), to reuse large-scale health data to address longstanding issues, such as those posed by SDH.

The use of health data warehouses (HDWs) offers an opportunity to collect and analyze accurate, real-world data, particularly through AI and NLP to extract information from medical reports. However, various challenges limit the use of NLP models, notably the dominance of models trained on English medical texts and privacy-related legislative restrictions. Therefore, alongside leveraging these models for clinical research, it is essential to continue efforts to develop transparent French-language models that comply with legislation.

Thus, the ARAMISS project proposes to study the interaction between SDH and known risk factors for IA rupture by comparing control populations and rupture cases. This study will be based on a certified health data warehouse (HDW) and an NLP algorithm previously developed by the team.

In parallel, the project plans two FAIR-compliant knowledge-sharing approaches to disseminate the algorithm and training corpus to the broader community.

DETAILED DESCRIPTION:
Intracranial aneurysms (IA), the most common intracranial arterial malformation, affect approximately 3% of the global population. They are characterized by a dilation of the vascular wall within the intracranial region, typically at a bifurcation. The most feared complication of IA is rupture, which is associated with high morbidity and mortality. About 30% of patients face death or severe disability, and even among those with no visible sequelae, up to 50% suffer from invisible disabilities such as cognitive problems. This explains the significant economic burden of ruptured IAs, estimated at approximately £168 million annually in the UK.

One way to reduce this morbidity and societal burden is to identify patients at high risk of rupture to determine those most likely to experience disease progression. Various initiatives, such as the ELAPSS, PHASES, and UCAS scores, have been developed to assess rupture risk in routine clinical practice. However, these scores largely rely on well-known modifiable and non-modifiable risk factors, such as ethnicity, hypertension, sex, age, smoking, and history of subarachnoid hemorrhage. Despite their utility, they are insufficient for reliably stratifying rupture risk, underestimating it by approximately 30%, which limits their impact in daily practice.

Recent research has identified emerging risk and protective factors, such as sleep apnea syndrome, lipid control, and the use of antidiabetic, lipid-lowering, or antihypertensive treatments. Therefore, it is necessary to revisit IA rupture risk by considering these factors in relation to patients' living environments.

Social determinants of health (SDOH) play a critical role in this context. Defined as the conditions of life that influence individual and population health, SDOH include broad factors such as age, ethnicity, and gender, as well as addiction behaviors, income levels, environmental exposure, and social status. They are estimated to contribute to over 80% of the population's health outcomes. In vascular diseases, SDOH -such as low education levels, limited income, social isolation, and low physical activity-are known to impact disease severity beyond traditional risk factors. The WHO estimates that vascular diseases are the leading global cause of mortality, with 17.7 million deaths annually, half of which are preventable. Understanding and addressing SDOH is therefore crucial for public health prevention efforts.

Initial studies on the impact of SDOH on IA rupture are limited, often focusing on individual determinants. A more comprehensive approach to SDH is needed, especially given the lack of consensus guidelines for IA management. Current therapeutic options, while advanced, still carry perioperative morbidity. Multivariable modeling and weighted composite scores can help address the complexity of clinical and environmental factors.

SDH data are routinely collected in medical records and increasingly digitized through hospital information systems. Health data warehouses (HDWs), such as the one at Nantes University Hospital, integrate structured and unstructured data from millions of patients, enabling their reuse for research purposes. The advent of artificial intelligence (AI) has made it possible to extract and analyze this data, revealing insights from previously inaccessible information.

Natural language processing (NLP), a branch of AI, enables automated extraction of information from textual medical records, unlocking the potential of unstructured data within HDWs. State-of-the-art models, such as BERT, ChatGPT, Llama, and Mistral, can process and analyze large volumes of text. However, the application of NLP to non-English languages is constrained by a lack of annotated corpora, privacy concerns, and data sovereignty regulations.

The ARAMISS project aims to investigate the interaction between SDH and known risk factors for IA rupture, comparing patients with unruptured IAs to those with ruptured IAs. Using SDH, the project will classify patients into risk groups and spatially analyze patient data through APIs like DataGouv. Additionally, the project will focus on developing FAIR (Findable, Accessible, Interoperable, Reusable) methodologies to share its algorithms and training corpora with the biomedical community while maintaining regulatory compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older at the time of their first cerebral imaging report mentioning an intracranial aneurysm (IA);
* Patients with a confirmed saccular IA based on imaging;
* Presence of at least one document referencing social determinants of health, lifestyle, habits, or exposure.

Exclusion Criteria:

* Patients who refuse the reuse of their health data;
* Patients diagnosed with dominant autosomal polycystic liver-kidney disease, sickle cell disease, mycotic aneurysm, fusiform aneurysm, blister-like aneurysm, Marfan syndrome, or Ehlers-Danlos syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Nantes Hospital aged 18 years or older at the time of their first cerebral imaging report mentioning an intracranial aneurysm (IA); with a confirmed saccular IA based on imaging.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Study the interaction between social determinants of health (SDH) and individual factors associated with intracranial aneurysm (IA) rupture using data available in the Nantes University Hospital Data Warehouse (EDS) | 18 months
  Calculate the Odds Ratios (OR) of explanatory factors related to the rupture outcome variable.

SECONDARY OUTCOMES:
Evaluate the impact of new risk factors on rupture occurrence | 18 months
  Evaluate the impact of new risk factors on rupture occurrence
  * Odds-Ratio for explanatory factors of the outcome variable, rupture. Demonstrate the protective effect of antihypertensive treatments on rupture risk
  * OR for explanatory factors of the outcome variable, rupture. Classify patients into homogeneous subgroups of individuals exposed to SDH
  * Subgroups. Classify patients spatially into geographical subgroups of rupture
  * Subgroup. Describe factors of social inequality influencing IA rupture occurrence
  * Percentage of prior healthcare access. Comment on Article 29 on data protection (GPDR)
  * White paper on data anonymity. Evaluate patient reidentification through language encoder models (BERT-type model)
  * Reidentification percentage. Compare the reidentifying characteristics of two language model training methods: models trained on entire de-identified documents vs. models trained on isolated de-identified sentences
  * Statistical significance of the difference.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes Hospital, Nantes, France, France